CLINICAL TRIAL: NCT07186192
Title: Digital Health Intervention for Self-Management and Telemonitoring in Chimeric Antigen Receptor-T Cell (CAR-T)Therapy
Brief Title: Digital Health Intervention for Self-Management and Telemonitoring in Chimeric Antigen Receptor (CAR-T) Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25328
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
Keywords: CAR-T; Digital health intervention
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - self-management coaching, telemonitoring (Experimental): Patients and their FCGs participate in self-management coaching sessions over 60 minutes each prior to CAR-T infusion and at approximately days 21, 42, and 70 post-CAR-T infusion. Beginning 15-20 days post CAR-T infusion, participants wear a FitBit device and use a mobile app QD three times per week for 90 days for tracking by nurses of daily steps, temperature, blood pressure, oxygen level, weight, and distress levels.
  Interventions: Other: Educational Intervention; Procedure: Health Telemonitoring; Other: Questionnaire Administration
- Arm B - Standard of Care Arm ( Enhanced usual care) (Active Comparator): Patients and their FCGs receive usual care, including standard print educational materials on study.
  Interventions: Other: Questionnaire Administration; Other: Best Practice

INTERVENTIONS:
Other: Educational Intervention — Patients and family caregivers that are randomized into the intervetnion arm (Digital health intervention) will receive a 90 day nurse-drive, digital health intervention. Participate in self-management coaching sessions
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
  Arms: Arm A - self-management coaching, telemonitoring
Procedure: Health Telemonitoring — Wear a FitBit device and use a mobile app for nurse tracking
  Arms: Arm A - self-management coaching, telemonitoring
Other: Questionnaire Administration — Ancillary studies
Other: Best Practice — Given usual care
  Other Names: best practice, standard of care, standard of care, standard of care, standard therapy
  Arms: Arm B - Standard of Care Arm ( Enhanced usual care)

SUMMARY:
The overall purpose of this randomized control trial (RCT) is to determine the clinical effect of a multilevel, RPM-enhanced intervention during and after completion of outpatient CAR-T therapy in 190 patients and their family caregivers (FCGs).

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria Informed Consent and Willingness to Participate

1. Documented informed consent of the participant and/or legally authorized representative Age and Language Criteria
2. Age ≥ 18 years old at the time of enrollment
3. Ability to read and understand English or Spanish for Questionnaires Nature of Illness and Treatment Related Criteria
4. Relapsed or refractory hematologic malignancy
5. Scheduled to receive outpatient standard of care (SOC) CAR-T therapy
6. Has a FCG committed to living with the patient for the duration of the study

Family Caregiver Inclusion Criteria Informed Consent and Willingness to Participate

1. Documented informed consent of the participant and/or legally authorized representative Age and Language Criteria
2. Age ≥ 18 years old at the time of enrollment
3. Ability to read and understand English or Spanish for Questionnaires Nature of Illness and Treatment Related Criteria
4. Family member or friend identified by the patient and defined as a person who knows the patient well and is involved in the patient's medical care

Exclusion Criteria 1. An employee who is under the direct/indirect supervision of the PI/ a co-investigator/ the study manager 2. A direct study team member

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2029-03-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory CAR-T module (MDASI-CAR - patient) | Baseline, Day 15 - Day 20 post-CAR-T, Day 30, Day 60, and Day 90
  This is validated measure of 22 CAR-T specific symptoms and other cancer-related symptoms. Symptom severity is rated on a 10-point scale: 1-3 mild, 4-6 moderate, ≥7 severe. Patients also rate how much their symptoms interfere with 6 functional domains: walking, activity, working/housework, relationships, enjoyment of life, and mood. A change in 1.2 points is clinically meaningful and cutoffs for clinical deficits have been defined. Cronbach's α reliability: 82-0.94.
Distress Thermometer (DT - FCG) | Baseline, Day 15 - Day 20 post-CAR-T, Day 30, Day 60, and Day 90
  This is an efficient, low-subject-burden measure to evaluate psychological distress over the past week, based on a scale of 0 (no distress) to 10 (extremely distressed). A cut-off of 3/10 indicates a need for intervention, with acceptable sensitivity (94.1%) and specificity (71.2%) compared to the longer Hospital Anxiety and Depression Scale (HADS). The DT has been validated in FCGs, and we chose it for its brevity, accuracy ease of use in remote monitoring, and validity in FCGs.

SECONDARY OUTCOMES:
Montgomery Borgatta Caregiver Burden Scale (FCG) | Baseline, Day 30, Day 60, and Day 90
  This is a 14-item tool designed to measure the impact of caregiving on three dimensions of burden: objective, subjective demand, and subjective stress. Internal consistency for the three dimensions ranges from 0.81-0.90. The ordinal scale ranges from 1-5 (a lot less to a lot more). The following cutoff scores are interpreted as high burden: 1) a score of ≥23 for objective burden, 2) a score of ≥15 for subjective demand, and 3) a score of ≥13.5 for subjective stress.
Functional Assessment of Cancer Therapy-General (FACTG - patient) | Baseline, Day 30, Day 60, and Day 90
  This is a cancer-specific version of the FACIT (Functional Assessment of Chronic Illness Therapy) Measurement System. It contains a 27-item compilation of general questions divided into four QoL domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. For each item, the respondent indicates on a 5-point Likert scale (0=not at all; 4=very much) how true each statement is for him/her during the past 7d. The FACT-G yields a total score for overall QoL as well as subscale scores. Internal consistency and reliability measures revealed a Cronbach's α of 0.89 for the total FACT-G, and a range of 0.70-0.82 for the four subscales.

OTHER OUTCOMES:
COH-QoL-Family (FCG) | Baseline, Day 30, Day 60, and Day 90
  This is a 37-item instrument that measures FCG QoL in the physical, psychological, social, and spiritual well-being domains. Ordinal scale ranges from 0-10, with higher scores indicating better QoL. The instrument was revised and tested from 1994-1998 in a study of 219 FCGs of cancer patients. The test-retest reliability was r=0.89 and internal consistency was α r=0.69.
Brief Dyadic Adjustment Scale (DAS - patient, FCG) | Baseline, Day 30, Day 60, and Day 90
  This is a 4-item scale designed to assess marital satisfaction for couples married or in a committed relationship. This instrument measures patient/FCG consensus, satisfaction, affectional expression and cohesion that directly assess general communication between couples. Alpha coefficients have been reported from 0.92 to 0.95. The measure will be included as a covariate for analysis. will be used to assess marital satisfaction (Patient, FCG).
FCG Activation in Transitions Tool (FCAT - FCG) | Baseline, Day 30, Day 60, and Day 90
  This is a 10-item survey designed to assess FCG's level of engagement and preparedness to care for patients during care transitions. Psychometric assessment was conducted in two randomly equivalent waves of participants (N=434), including FCGs of patients with cancer and/or chronic lung disease. The estimated person-separation reliability was 0.84.
Patient Activation Measure (PAM - patient) | Baseline, Day 30, Day 60, and Day 90
  This is a measure of patient "activation", which uses a Guttman-like scale that reflects patient level of engagement and empowerment in their healthcare. Cronbach's α from our pilot study was 0.92.
PROMIS Self-Efficacy for Managing Symptoms Short Forms 8a (patient) | Baseline, Day 30, Day 60, and Day 90
  This is a brief, 8-item questionnaire used to assess an individual's confidence in their ability to manage specific aspects of symptoms. Specifically, the tool measures confidence in managing symptoms during daily activities, social interactions, and in public places.
Self-Efficacy Scale (FCG) | Baseline, Day 30, Day 60, and Day 90
  This is a modified version of the Self-Efficacy Scale. Contains 8 items that assess FCG perceived confidence in self-management. Uses a 4-point Likert scale; higher scores represent greater confidence. Cronbach's α from our pilot: 0.89.
Sociodemographic and Health Status (patient) | Baseline
  This is a questionnaire to assess patient demographics.
FCG Demographics (FCG) | Baseline
  This is a questionnaire to assess patient demographics.
Acceptability of Intervention (AIM) - Acceptability | Patients: Day 90 only; CAR-T clinical care team: before intervention starts and after intervention ends
  This is a questionnaire used to assess patient, family caregiver, and CAR-T clinical care team on acceptability of the intervention.
Intervention Appropriateness Measure (IAM) - Appropriateness | Patients: Day 90 only; CAR-T clinical care team: before intervention starts and after intervention ends
  This is a questionnaire used to assess patient, family caregiver, and CAR-T clinical care team on the appropriateness of the intervention.
Feasibility of Intervention (FIM) | Patients: Day 90 only; CAR-T clinical care team: before intervention starts and after intervention ends
  This is a questionnaire used to assess patient, family caregiver, and CAR-T clinical care team on the feasibility of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, PhD, RN, Principal Investigator — City of Hope Medical Center; Saro Armenian, DO, MPH, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided